CLINICAL TRIAL: NCT05683223
Title: Neural Markers of Treatment Mechanisms and Prediction of Treatment Outcomes in Social Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Massachusetts Institute of Technology (Other); Mclean Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anthony J. Rosellini, Associate Professor, Boston University Charles River Campus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH128377 (NIH); R01MH128377 (NIH)
Record Dates: First submitted 2022-12-19; First posted 2023-01-13 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Social Anxiety Disorder
Keywords: social anxiety disorder; sertraline; exposure therapy; social cost; MRI; EEG; structural connectivity; functional connectivity; cognitive control system; positive valence system; negative valence system
MeSH Terms: conditions — Phobia, Social | interventions — Sertraline

STUDY DESIGN:
Intervention Model Description: 1. Recruit 240 participants, with 190 meeting criteria for SAD and 50 serving as non-psychiatric controls;
  2. Treat 190 SAD patients with CBT for SAD, and treat nonresponders with CBT plus SSRI;
Masking Description: N/A--no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Responders (Experimental): The experimental arm involves EEG + MRI before and after exposure therapy for social anxiety disorder.
  Interventions: Behavioral: Group CBT for Social Anxiety Disorder
- Non-Responders (Experimental): The experimental arm involves EEG + MRI before and after exposure therapy for social anxiety disorder. Non-responders to initial exposure therapy will receive sertraline and additional exposure therapy prior to final EEG and MRI.
  Interventions: Behavioral: Group CBT for Social Anxiety Disorder; Drug: Sertraline; Behavioral: Individual CBT for Social Anxiety Disorder
- Controls (No Intervention): Controls will receive baseline EEG and MRI, screening questionnaires and intake interview. They will not participate in therapy but complete weekly symptom measures and a second EEG/MRI session 12 weeks after baseline. Control participants will be compared with social anxiety participants to determine differences in neuro-markers at baseline and over follow-up.

INTERVENTIONS:
Behavioral: Group CBT for Social Anxiety Disorder — Initial CBT will consist of 12 weekly, 2.5-hour group sessions. Later sessions (after session 7) become more individualized as the exposure practices are tailored to the individual participant's concerns. Most often, the exposures are completed outside the group environment. Session content includes various cognitive behavioral strategies tailored to SAD, such as psychoeducation, examining and challenging cognitive distortions, and exposure exercises.
  Other Names: SAD Group
  Arms: Non-Responders; Responders
Drug: Sertraline — Non-responders will initiate sertraline at baseline (week 0) with 25 mg/day followed by a dose increase to 50 mg/day at week 1, 100 mg at week 4, 150 mg at week 6, and 200 mg at week 8. Upward dose titration may be slowed and the dose decreased if necessary due to side effects, but the clinician will attempt to titrate all symptomatic participants up to 200 mg/day if tolerated by week 8, with the last dose increase allowed at week 10. Participants will be assessed at each visit by the study psychiatrist for purposes of dose titration and monitoring. Symptomatic participants unable to reach 200 mg/day of sertraline due to side effects will be maintained in the trial if they are on at least 50 mg/day by week 8; all symptomatic participants will be titrated to their maximally tolerated dose (< 200 mg/day sertraline). Any participant unable to tolerate sertraline will be discontinued and referred for clinical treatment.
  Other Names: Non-responder Meds
  Arms: Non-Responders
Behavioral: Individual CBT for Social Anxiety Disorder — Participants who show no or only partial response to the initial group CBT will continue with an individual, tailored form of CBT plus adjunctive SSRI. The format of CBT will include
  Other Names: Non-responder CBT
  Arms: Non-Responders

SUMMARY:
The purpose of this clinical trial is to answer the question: can the investigators predict which adults with social anxiety disorder (SAD) will successfully respond to treatment? To answer this question, the investigators plan to recruit 190 adult participants who experience extreme forms of social anxiety to undergo brain imaging before and after 12 weeks of group cognitive behavioral therapy (CBT). Adults in the SAD group who do not respond enough to group CBT may be offered the opportunity to complete an additional 12 weeks of individual CBT while receiving SSRI medication (sertraline, see below) for SAD.

Data collected from participants who experience anxiety will be compared to a group of 50 participants with little or no social anxiety, who will serve as a comparison group.

DETAILED DESCRIPTION:
The primary aim of this study is to discover neural mechanisms (via EEG and MRI) associated with variation in response to CBT and/or combined CBT and SSRI interventions. The goal is to develop a rigorous model that predicts individual differences in response to treatments using baseline neural markers.

The investigators will recruit 190 adults with social anxiety disorder (SAD) and 50 adult controls. All adults with SAD will participate in group CBT for SAD. Non-responders will continue on with individual CBT plus the addition of sertraline for another 12 weeks. 50 controls will receive baseline EEG and MRI but will not participate in any clinical interventions. The investigators will also perform neuroimaging (task fMRI, rsfMRI, DWI, structural MRI) and collect EEG before treatment, to compare patient and control groups, and to obtain neuromarkers that predict treatment response.

MRI/EEG Tasks

Activation of Negative Valence System. The RDoC recommends "viewing aversive pictures" as a means to activate the Negative Valence System. The investigators will adapt the paradigm that accounted for 40% of CBT outcome variance in which participants viewed blocks of angry or neutral faces. The investigators chose to use a block (rather than an event-related) design because block designs have stronger measurement power for characterizing individuals. Experimental design. Stimuli will be color faces from the NimStim set with angry or neutral expressions. There will be six 15-second blocks per condition, with six faces per block; each face is presented for 1250 ms, followed by 1250 ms of fixation. The task starts and ends with a fixation block, and each pair of face blocks is separated by one fixation block. Two fixed forms are used to counterbalance condition orders. Participants perform a 1-back task by indicating, via button press, the repetition of a face.

Activation of Positive Valence System. As reviewed in Significance, there is evidence that the reward system is atypical in SAD. To investigate this further, the investigators will adapt a widely used reward processing task that was developed by Delgado and that is recommended by the RDoC for probing the initial response to reward. Experimental design. Participants play a guessing game to try to win money. Each trial begins with presentation of a "mystery card" displaying a "?" (duration: 1.5s). Participants are told that card numbers range from 1 to 9, and they indicate whether they think the mystery card number on a given trial is more or less than 5 by pressing a button. Feedback (1s) is given immediately after and consists of either (a) a reward (a green up arrow and "$1"), (b) a loss (red down arrow with "-$0.50"), or (c) a neutral outcome (the number 5 and a grey double-headed arrow). A 1 s intertrial interval (ITI) separates the trials. Participants complete two runs, each of which includes four blocks of eight trials: two blocks yield mostly rewards (6/8 trials), and two blocks yield mostly losses (6/8 trials). There are also four 15 s fixations, to facilitate deconvolution of fMRI responses.

Activation of Cognitive Control System. Based on encouraging prior findings, the investigators have included a cognitive control task in which pretreatment activation of dorsal anterior cingulate cortex (dACC) predicted response to CBT+SSRI in SAD with 83% accuracy. Experimental design. The task is known as the MSIT. It has four blocks each of two conditions (control and interference). Each block lasts 42 s and consists of 24 trials (1750 ms per trial) in pseudo-randomized order with sets of 3 digits (0, 1, 2, or 3) centrally displayed. One "target" digit differs from the other two (distractors). In the control condition, the distractors are always '0' and the target digit corresponds to its position (i.e., '1' in the leftmost position; '2' in the middle position; and '3' in the rightmost position). Thus, on control trials, the target digit and position are congruent. In the interference condition, the distractors are '1', '2', or '3' and the target digit and position are incongruent (e.g., '1' presented in the rightmost position). Participants indicate if the target digit is '1', '2', or '3' by pressing the response buttons. Ignoring the distractors and the misleading position of the target digit on interference trials requires cognitive control.

Our primary hypotheses are that: (1) The investigators will identify patterns of brain activity that distinguish adults with SAD from adults in the comparison group, and that (2) The investigators will be able to identify patterns of brain activity that predict which adults with SAD will (or will not) respond to treatment.

The primary outcome measure will be treatment response (defined elsewhere in this registration).

ELIGIBILITY:
Inclusion criteria for all participants:

(1) Any gender or race between 18-50 years old.

Additional inclusion criteria for healthy controls:

(1) Liebowitz Social Anxiety Scale (LSAS; Mennin et al., 2002) score <= 30, does not currently meet criteria for an Axis I psychiatric condition, as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5; American Psychiatric Association, 2013).

Additional inclusion criteria for the social anxiety disorder (SAD) group:

1. Outpatients with a primary psychiatric complaint (designated by the patient as the most important source of current distress) of social anxiety with social interaction fear as defined by an Liebowitz Social Anxiety Scale (LSAS) score >= 60.
2. Overall clinical severity of at least mild as defined by Clinical Global Impressions Scale (CGI-S; Zaider et al., 2003) of at least 3.
3. Medical history interview and laboratory findings without clinically significant abnormalities.
4. Willingness and ability to participate in the informed consent process and comply with the requirements of the study protocol.

Exclusion criteria:

1. A lifetime history of bipolar disorder, schizophrenia, psychosis, delusional disorders or obsessive-compulsive disorder; an eating disorder in the past 6 months; organic brain syndrome, intellectual disability, or other cognitive dysfunction that could interfere with capacity to engage in therapy; a history of substance or alcohol abuse or dependence (other than nicotine) in the last 6 months or otherwise unable to commit to refraining from alcohol, marijuana, and stimulant use during the acute period of study participation.
2. . Patients with significant suicidal ideation Montgomery-Åsberg Depression Rating Scale (10 items, self-report) or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
3. Patients can be taking a concurrent psychotropic medication (e.g., antidepressants, anxiolytics, beta blockers, sertraline), but the dose must be stabilized for at least 2 weeks prior to initiation of randomized treatment.
4. Significant personality dysfunction likely to interfere with study participation.
5. Serious medical illness, associated treatment, or other instability for which hospitalization may be likely within the next year, or which may alter fMRI or EEG measurements. Participants with a history of serious medical illness or treatments that may alter fMRI measurements may enroll in the study 12 months after the condition has been remitted and ending treatment.
6. Patients with a current or past history of seizures.
7. Pregnant women, lactating women, and women of childbearing potential who may become pregnant.
8. Any concurrent psychotherapy initiated within 3 months of baseline, or ongoing psychotherapy of any duration directed specifically toward treatment of the social anxiety is excluded. Individuals with prior CBT experience or treatments that included cognitive and behavioral skills and exposure procedures (e.g., assertiveness and social skills trainings) will be excluded. General supportive or insight-oriented therapy initiated > 3 months prior is acceptable.
9. Prior non-response to adequately-delivered exposure (i.e., as defined by the patient's report of receiving specific and regular exposure assignments as part of a previous treatment).
10. Patients with a history of head trauma causing loss of consciousness, seizure or ongoing cognitive impairment.
11. Contraindications for MRI including metal implants, surgical clips, probability of metal fragments, braces, or claustrophobia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Global Impression-Improvement Scale (CGI-I) | 6 weeks, 12 weeks, 19 and 25 weeks for non-responders
  The CGI-S is a 7-point scale that requires the clinician to rate the improvement of the patient's illness at the time of assessment compared to baseline. To aid CGI scoring, the clinician will use the Social Phobic Disorders Severity and Change Form (SPD-SC). Treatment responder status will be defined as a CGI-I score of 1 (very much improved) or 2 (much improved)
Change in Liebowitz Social Anxiety Scale (LSAS) | Before Week 0, 6 weeks, 12 weeks, 19 and 25 weeks for non-responders
  The LSAS is a questionnaire developed by Dr. Michael R. Liebowitz, a psychiatrist and researcher. This measure assesses the way that social phobia plays a role in the participant's life across a variety of situations. LSAS greater than or equal to 60 meets criteria for inclusion in the treatment group.

SECONDARY OUTCOMES:
Change in Clinical Global Impression Severity scale (CGI-S) | Week 0, 6 weeks, 12 weeks, 19 and 25 weeks for non-responders
  The CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Ratings range from 1 (normal) to 7 (most extremely ill patients). CGI-S greater than or equal to 3 meets criteria for inclusion in SAD treatment group.
Social Phobia Inventory (SPIN) | Weekly up through week 12, and weekly from weeks 14-25
  The Social Phobia Inventory (abbreviated as SPIN ) is a 17-item questionnaire developed by the Psychiatry and Behavioral Sciences Department at Duke University. Each item is rated 0 (not at all) to 4 (extremely). It is effective in screening for, and measuring the severity of social anxiety disorder.
The Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) | Week 0, 6 weeks, 12 weeks, 19 and 25 weeks for non-responders
  The Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) is a 16-item self-report measure designed to enable investigators to easily obtain sensitive measures of the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning. The measure rates aspects of quality of life, including physical health, mood, activities of daily living, and overall life satisfaction on a scale from 1 (very poor) to 5 (very good).
Social Network Index (SNI) | Week 0, 6 weeks, 12 weeks, 19 and 25 weeks for non-responders
  The 12-item SNI questionnaire assesses 12 types of social relationships. This measure will be included in secondary exploratory analyses as a baseline measure for change with treatment. Assessment scores are summed with 0 being the most isolated, and 2, 3, and 4 forming categorizations of increasing social connectedness.
Patient Health Questionnaire-9 (PHQ-9) | Weekly up through week 12, and weekly from weeks 14-25
  The PHQ-9 is a nine-item diagnostic self-report questionnaire which psychologists use to measure the severity of depressive symptoms in patients with mood disorders. This measure will be used to monitor weekly depression symptoms, and scores greater than or equal to 4 indicate clinical levels of depression. Each item is scored on a scale of 0 to 3, with 0 indicating "not at all" and 3 denoting "present nearly every day". The total score range is 0-27.
General Anxiety Disorder-7 (GAD-7) | Week 0, 6 weeks, 12 weeks, 19 and 25 weeks for non-responders
  The GAD-7 is a seven-item diagnostic self-report questionnaire which psychologists use to measure the severity of anxiety symptoms in patients with mood disorders. This measure will be used to monitor weekly anxiety symptoms, and scores greater than or equal to 5 indicate clinical levels of anxiety. Each item is scored on a scale of 0 to 3, with 0 meaning "not at all" and 3 denoting "present nearly every day". The total score range is 0-21.
Social Anxiety Questionnaire (SAQ) | Week 0, 6 weeks, 12 weeks, 19 and 25 weeks for non-responders
  The SAQ is a 30-item measure of social anxiety consisting of 30 items and five subscales. Each item is rated on a 5-point scale, with a high score indicating a higher social anxiety level.
Changes in the Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders (DIAMOND) | Week 0, 6 weeks, 12 weeks, 19 and 25 weeks for non-responders
  The DIAMOND is a semi-structured interview guide for making the major DSM-5 diagnoses. It is administered by a clinician or trained mental health professional who is familiar with the DSM-5 classification and diagnostic criteria. This measure will be used to determine eligibility for the study in conjunction with other primary outcome measures.

OTHER OUTCOMES:
Social Cost Questionnaire (SCQ) | Week 0, 6 weeks, 12 weeks, 19 and 25 weeks for non-responders
  The SCQ is a 40-item measure that examines a person's assessment of the negative consequences of a social mishap. Each item is scored 0 (not at all) to 8 (extremely). We will administer this questionnaire at each session to examine whether it differentially mediates change with CBT vs. pharmacotherapy.
Kaufman Brief Intelligence Test (KBIT) | Week 0
  The Kaufman Brief Intelligence Test is used to measure verbal and non-verbal intelligence in individuals from ages 4 through 90 years. This measure will be administered at baseline for consideration as a potential moderator of treatment response. Verbal and non-verbal scales are finally scored, standardized for age, and are able to be transformed into an IQ score with a mean of 100 and standard deviation of 15. Overall scores range from 40 to 160, with higher scores indicating a better outcome.
Credibility/Expectancy Questionnaire (CEQ) | Week 0
  The Credibility/Expectancy Questionnaire is the most widely used measure of treatment credibility and expectancy in psychotherapy research. This measure will be administered at baseline as a potential moderator of treatment response. This questionnaire utilizes two scales, 1-9 and 0-100%, with higher scores meaning a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: John Gabrieli, PhD, Principal Investigator — Massachusetts Institute of Technology; Daniel Dillon, PhD, Principal Investigator — Mclean Hospital; Anthony Rosellini, PhD, Principal Investigator — Boston University Charles River Campus
Locations (1):
- Center for Anxiety and Related Disorders at Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
REDCap will create appropriately de-identified databases according to guidelines provided by the NIH and research data sharing practices. A de-identified dataset can be readily shared without the need of a Data Use Agreement (DUA) and facilitates book-keeping, making it the preferred data sharing plan. All study data will be made available via a data archive accessible through a public website hosted by McLean, BU, and/or MIT. Web archived data may also be available as downloadable content. Our data sharing policies and capabilities will follow published NIH standards relating to data sharing. Access to databases generated under the project will be available for educational, research and non-profit purposes. Such access will be provided using web-based applications, as appropriate.
  Further, all de-identified data will be shared with appropriate permissions with the National Database for Clinical Trials related to Mental Illness (NDCT), and thus available for all researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: In accordance with NIMH policies, these data will be made available within twelve months of database lock or following publication of primary manuscript, whichever occurs first.
Access Criteria: Access criteria will align with requirements for access to NDCT and other NIMH databases.

REFERENCES:
- [Background] Bush G, Shin LM, Holmes J, Rosen BR, Vogt BA. The Multi-Source Interference Task: validation study with fMRI in individual subjects. Mol Psychiatry. 2003 Jan;8(1):60-70. doi: 10.1038/sj.mp.4001217. PMID 12556909
- [Background] Delgado MR, Nystrom LE, Fissell C, Noll DC, Fiez JA. Tracking the hemodynamic responses to reward and punishment in the striatum. J Neurophysiol. 2000 Dec;84(6):3072-7. doi: 10.1152/jn.2000.84.6.3072. PMID 11110834
- [Background] Tottenham N, Tanaka JW, Leon AC, McCarry T, Nurse M, Hare TA, Marcus DJ, Westerlund A, Casey BJ, Nelson C. The NimStim set of facial expressions: judgments from untrained research participants. Psychiatry Res. 2009 Aug 15;168(3):242-9. doi: 10.1016/j.psychres.2008.05.006. Epub 2009 Jun 28. PMID 19564050